CLINICAL TRIAL: NCT00478426
Title: A Phase 2 Study of Sunitinib Malate in Recurrent or Metastatic Endometrial Carcinoma
Brief Title: Sunitinib Malate in Treating Patients With Recurrent or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00210; NCI-2009-00210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-062; CDR0000513153; 7713 (Other: University Health Network-Princess Margaret Hospital); 7713 (Other: CTEP); N01CM62201 (NIH); N01CM62203 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Serous Adenocarcinoma; Recurrent Uterine Corpus Carcinoma; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7; Uterine Carcinosarcoma; Uterine Corpus Carcinosarcoma
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO QD on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies how well sunitinib malate works in treating patients with endometrial cancer that has come back after a period of improvement (recurrent) or has spread to other places in the body (metastatic). Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate of recurrent or metastatic endometrial cancer to sunitinib (sunitinib malate).

II. To assess the frequency of prolonged stable disease (as defined by percentage [%] of patients alive and free from progressive disease at 6 months) in patients with recurrent or metastatic endometrial cancer treated with sunitinib.

SECONDARY OBJECTIVES:

I. To assess time-to- progression, median overall survival, and rate of one-year survival in patients with recurrent or metastatic endometrial cancer treated with sunitinib.

II. To assess the toxicity associated with sunitinib in patients with recurrent or metastatic endometrial cancer.

OUTLINE:

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed up at 4 weeks and then every 3 months until relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed endometrial cancer; adenocarcinoma (endometrioid and serous/papillary serous) and carcinosarcoma (ie. malignant mixed Mullerian tumor [MMMT]) of the uterus will be investigated; patients with other histologies (eg. squamous cell carcinoma or leiomyosarcoma) are excluded
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; indicator lesions must not have been previously treated with surgery, radiotherapy, or radiofrequency ablation
* Previously treated patients must have evidence of progressive disease, either clinically or radiographically, as assessed by the investigator
* Eligible patients may have received no more than one prior cytotoxic chemotherapy regimen for recurrent, locally-advanced, or metastatic disease; if the prior chemotherapy was an anthracycline, they may have received no more than 6 cycles (or less than 450 mg/m^2 doxorubicin); patients must have completed any previous chemotherapy a minimum of 4 weeks (or 6 weeks if the regimen contained carmustine [BCNU] or mitomycin) prior to study registration; prior investigational treatment is permissible (as long as such treatment completed 4 weeks prior to registration)
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 100 g/dL
* Serum calcium =< 12.0 mg/dL (=< 3.0 mmol/L)
* Total serum bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Serum lipase =< 1.5 x institutional upper limit of normal
* Serum amylase =< 1.5 x institutional upper limit of normal
* Thyroid stimulating hormone (TSH)/T3/T4 within normal institutional limits
* Magnesium >= 0.5 mmol/L
* Patients must have corrected QT interval (QTc) < 500 msec
* The following group of patients are eligible provided they have normal baseline cardiac function (as determined by estimate of left ventricular ejection fraction [LVEF] on echocardiogram or multi-gated acquisition scan [MUGA]):

  * Those with a history of congestive heart failure, provided they are no greater than New York Heart Association (NYHA) class I and on treatment at baseline
  * Those with prior anthracycline exposure
  * Those who have received prior central thoracic radiation that included the heart in the radiotherapy port
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; all women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; at least 4 weeks must have elapsed since any major surgery
* Patients may not be receiving any other investigational agents
* Patients who have received prior treatment with any other antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, PTK787, vascular endothelial growth factor [VEGF] Trap, etc.) are ineligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib
* Patients who have a history of serious ventricular arrhythmias (ventricular tachycardia [VT] or ventricular fibrillation [VF] equal to or greater than 3 beats in a row), QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities are excluded
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) are ineligible
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: Low molecular weight heparin is permitted provided the patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
  * Class III or IV heart failure as defined by the NYHA functional classification system
  * Pre-existing adrenal insufficiency (primary or secondary)
* The eligibility of patients taking medications that are potent inducers or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) will be determined following a review of their case by the Principal Investigator; every effort should be made to switch patients taking such agents or substances to other medications, particularly patients who are taking enzyme-inducing anticonvulsant agents
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible
* Patients with known brain metastases should be excluded
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with sunitinib malate
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Oza, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (29):
- United States (21):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Evanston Hospital CCOP, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Result] Castonguay V, Lheureux S, Welch S, Mackay HJ, Hirte H, Fleming G, Morgan R, Wang L, Blattler C, Ivy PS, Oza AM. A phase II trial of sunitinib in women with metastatic or recurrent endometrial carcinoma: a study of the Princess Margaret, Chicago and California Consortia. Gynecol Oncol. 2014 Aug;134(2):274-80. doi: 10.1016/j.ygyno.2014.05.016. Epub 2014 May 29. PMID 24882554

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sunitinib Malate)
Started | 34
Completed | 33
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 34 women with with endometrial cancer (subtypes included endometrioid, serous and carcinosarcoma) were enrolled onto the study. One participant with endometroid endometrial cancer withdrew consent prior to treatment, resulting in 33 participants receiving at least one dose of the study drug and were thus considered eligible for analysis.
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 65 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 22
  United States | 12
Endometrioid Subtype [Count of Participants; unit: Participants] | 24
Serous Subtype [Count of Participants; unit: Participants] | 6
Carcinosarcoma Subtype [Count of Participants; unit: Participants] | 3
Number of Lines of Previous Therapies [Count of Participants; unit: Participants]
  0 prior lines of therapy | 9
  1 prior line of therapy | 17
  2 prior lines of therapy | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate, defined as the rate of complete or partial response as defined by the Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), disappearance of all target lesions.
Time Frame: Up to 7 years
Population: Of the 33 participants, only 28 were considered evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 33
Participants
  Partial Response | 6
  Stable Disease | 6
  Progressive Disease | 16
  non-evaluable patient | 5

2. Secondary Outcome: Number of Participants With Prolonged Stable Disease
Description: Described as the best response of stable disease that is maintained for atleast 6 months
Time Frame: Up to 7 years
Population: Of the 33 participants, 28 were considered evaluable for response. 5 of these patients were not fully evaluable for the study as they were removed before first radiological assessment but are nonetheless included in denominator for response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 33
Participants | 0

3. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.
Time Frame: Up to 7 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 33
months | 19.4 [6.2 to 60]

4. Secondary Outcome: Number of Participants With Adverse Effects Assessed by CTCAE Version 3.0
Description: Number of participants that experience at east 1 adverse event while on trial, according to the CTCAE.
Time Frame: Up to 7 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 33
Participants | 30

5. Secondary Outcome: Time to Progression
Description: The length of time from the date of diagnosis or the start of treatment for a disease until the disease starts to get worse or spread to other parts of the body. Assessed by Kaplan and Meier method
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 33
months | 3 [2.5 to 5.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline, onward to end of treatment up to 5 years total.
Arm/Group | Treatment (Sunitinib Malate)
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 30/33
Other Adverse Events (participants affected / at risk) | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sunitinib Malate) (N=33)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 14 (14)
Hypertension (Cardiac disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sunitinib Malate) (N=33)
Diarrhea (Gastrointestinal disorders) | 25 (25)
Dyspepsia (Gastrointestinal disorders) | 17 (17)
Oral Mucositis (General disorders) | 17 (17)
Nausea (Gastrointestinal disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT00478426/Prot_SAP_000.pdf